CLINICAL TRIAL: NCT07177261
Title: Inter-Brain Synchrony as a Neural Mechanism of Social Connection in Schizophrenia
Brief Title: Inter-Brain Synchrony in Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jonathan Wynn, PhD, Researcher, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-25-1279; 1R21MH139044-01A1 (NIH)
Record Dates: First submitted 2025-09-02; First posted 2025-09-16 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia Disorder
Keywords: schizophrenia; EEG; interbrain synchrony; hyperscanning; social connections
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast Friends (Experimental): Participants will interact with another person while both have their EEG recorded. Participants will ask and answer 12 questions with the other person that become increasingly personal in nature, e.g., "When did you last cry in front of another person? By yourself?"
  Interventions: Behavioral: Fast Friends
- Small Talk (Active Comparator): Participants will interact with another person while both have their EEG recorded. Participants will ask and answer 12 impersonal questions with the other person , e.g., "Do you prefer digital watches and clocks or the kind with hands? Why?"
  Interventions: Behavioral: Small Talk

INTERVENTIONS:
Behavioral: Fast Friends — Participants will interact with another person while both have their EEG recorded. They will ask and answer 12 questions with the other person that become increasingly personal in nature, e.g., "When did you last cry in front of another person? By yourself?"
  Arms: Fast Friends
Behavioral: Small Talk — Participants will interact with another person while both have their EEG recorded. They will ask and answer 12 impersonal questions with the other person , e.g., "Do you prefer digital watches and clocks or the kind with hands? Why?"
  Arms: Small Talk

SUMMARY:
The goal of this clinical trial is to investigate for the first time in people with schizophrenia a neural mechanism that is thought to facilitate the formation of social connections - inter-brain synchrony - in order to improve scientific understanding of the neural mechanisms of social dysfunction in the disorder, and to provide a basis for the development of new and better treatments to improve social functioning and connectedness in the illness. The main questions it aims to answer are:

1. Investigate inter-brain synchrony as a neural mechanism of social connection in schizophrenia
2. Manipulate social closeness and test for effects on inter-brain synchrony across groups

The investigators will compare results from people with schizophrenia to a healthy comparison group (controls) who do not have psychotic disorders to see if inter-brain synchrony is greater in controls. Investigators will also compare measures of inter-brain synchrony before and after the social closeness manipulation to see if inter-brain synchrony changes with increasing closeness.

Participants will:

* Have a clinicial diagnostic interview and be assessed for clinical symptoms
* Have an EEG recorded while interacting with another person. Participants will first work with the other person to draw a figure, and then tap fingers together. Participants will then either undergo the experimental manipulation to increase social closeness (called, "fast friends") or undergo the control condition that does not increase social closeness (called "small talk"). Participants will then repeat the drawing and finger tapping assessment.
* After completing the experimental or control condition, participants will then repeat the procedure with the other condition that was not yet done.
* Be interviewed on the number and quality of social interactions.

ELIGIBILITY:
Inclusion Criteria:

* sufficient English fluency to comprehend procedures
* clinical group will include individuals with a DSM-5 diagnosis of schizophrenia who are clinically stable (outpatients, with no hospitalizations 3 months prior to enrollment and no medication changes 1 month prior to enrollment)
* members of the community without a psychotic disorder, schizophrenia-spectrum disorder, or current major mood disorder, nor history of a first-degree relative with a psychotic disorder.

Exclusion Criteria:

* evidence of IQ < 70 or developmental disability
* history of significant neurological disease, serious head injury, or significant current substance use (moderate or severe substance use disorder in the last 3 months, positive urine toxicology screen on the day of assessment, or sedatives/anxiolytics taken within 12 hours of the assessment)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Interbrain synchrony | Interbrain synchrony will be measured immediately before and immediately following the procedure.
  Circular correlations for 8-10Hz activity across electrodes and dyads

SECONDARY OUTCOMES:
Social Network Analysis | Measured at the start of the study only
  Measures of social and family social connections. Participants will be interviewed about the number of social and family connections they have, and if these contacts also know others identified by the participant. These connections will be analyzed with graph network analyses to determine the size and quality of social connections.
Behavioral measures of synchrony | Investigators will measure these during each of the two maniuplations (small talk and fast friends).
  Investigators will video record interactions between dyads (including voice, body, face) and measure behavioral measures of synchrony

CONTACTS AND LOCATIONS:
Overall Officials: Eric Reavis, Phd, Principal Investigator — University of California, Los Angeles; Jonathan K Wynn, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
EEG measures of interbrain synchrony, clinicial symptom ratings, social connectedness measures
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: At the end of the study (November 2027) for indefinite period
Access Criteria: These data will be shared on the NIMH Data Archive